CLINICAL TRIAL: NCT05405140
Title: Multiphasic Neuroplasticity Based Training Protocol With Shock Wave Therapy For Post Stroke Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/1102
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Spasticity, Muscle
Keywords: Neuroplasticity,; Exercise; Stroke; post stroke spasticity; Electromyography; Ultrasonography
MeSH Terms: conditions — Stroke; Muscle Spasticity; Motor Activity | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shock wave therapy with multiphasic neuroplasticity based training protocol (Experimental): Shock wave therapy with multiphasic neuroplasticity based training protocol based on motor relearning program and task oriented approach
  Interventions: Other: Shock wave therapy with multiphasic neuroplasticity based training protocol
- Conventional physical therapy (Active Comparator): Stretching and strengthing and motor sensory motor training of effected side
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Shock wave therapy with multiphasic neuroplasticity based training protocol — Interventions program will be based on Activity dependent neuroplasticity targeting relevant impairments included: task specific practice, motor learning, strengthening, postural awareness, Balance training, aerobic and conditioning exercises, range of movement with Shock wave therapy for most of time of the day .
  Arms: Shock wave therapy with multiphasic neuroplasticity based training protocol
Other: Conventional physical therapy — The CP program focused on the facilitation of movements on the paretic side, range of motion, stretching exercises, upper and lower limb strengthening exercises, and improving balance, standing, sitting, transferring, patients received a program for at least 30 sessions, 5 times per week for 6 or more weeks.
  Arms: Conventional physical therapy

SUMMARY:
this study will be conducted to f find the effects of multiphasic neuroplasticity based training protocol with Shock Wave Therapy on Neurophysiological, Morphological and Functional Parameters of Post Stroke Spasticity.

DETAILED DESCRIPTION:
Spasticity is a common sensory-motor dysfunction observed following a stroke. Spasticity is a velocity-dependent increase in resistance during a passive stretch due to hyper excitability of stretch reflex. This results in many functional impairments and patients centered problems. Given the complexity of spasticity related issues, its rehabilitation must entail comprehensive approach which address and synchronize spasticity reduction with motor function restoration without compensation. Shock Wave Therapy (SWT) is a non-invasive low cost devise gaining its use for spasticity reduction. After damage brain undergoes some sort of rearrangement. Literature says that during this period if it will rehabilitated through new pattern functional recovery can be optimized. However there is paucity of evidence for effectiveness of multiphasic neuroplasticity based Training protocol (MNTP) with SWT regarding its intensity frequency and specificity for spasticity management.

It will be a mix method approach. The patients after full filling the inclusion criteria , age ranging between 45 to 65 years having a stroke more than 3 months ago and having problematic spasticity interfering with function or causing a clinical problem, and no contraindications to shock wave therapy Upper or lower limb spasticity MAS ≥ 1 will be randomly assigned into four groups A,B,C,D. All groups will receive conventional rehabilitation training for 30 min per day five times a week for 4 weeks .Moreover patients in group A,BC also receive added SWT, MNTP and a combination of MNTP and SWT respectively. Motor recovery and spasticity will be using clinical (modified Asworth scale, Tardieu scale), neurophysiological, morphological(muscle ultrasound) and functional parameter( Fugl -meyer, burg balance, time up and go, Barthal index, Rivermeads mobility index ) at 0 , 8 and 16 week of treatment. The methodological approach used in this, will encompasses quantitative methods to assess program effectiveness and mixed methods to evaluate rehabilitation program components and aspects of protocol implementation. Qualitative methodology is needed to capture the range of participant experiences in the real- life clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* 40 - 70years.

  * Those had a stroke more than 3 months ago
  * Unilateral stroke
  * Able to participate in therapy regime or Participate in an ambulatory rehabilitation program.
  * They having problematic spasticity either focal or generalized.
  * Upper or lower limb spasticity (MAS ≥ 2) interfering with function or causing a clinical problem, and no contraindications to shock wave therapy.
  * if the improvement in spasticity is realistically expected
  * they will be considered suitable for to shock wave therapy
  * Minimental scale examination (MMSE).
  * Comprehensive Severity Index (CSI) for severity assessment.

Exclusion Criteria:

* If they had had received treatment with BoNT-A within six months
* Will receiving intrathecal baclofen or other anti-spasticity medications
* If patients will be on to anticoagulants.
* had undergone neurolysis or surgery to the affected limb;
* had concomitant neurological conditions

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Modified ashworh scale | 6th weeks
  Modified Ashworth Scale (MAS) is used to assess spasticity. Scoring is between 0 to 4 where 0 means no increase in muscle tone and 4 means limb is rigid in flexion or extension.

SECONDARY OUTCOMES:
Resting joint angle | 6th weeks
  Resting joint angle will showa the spasticity, the most the angle is narrow the more the mucle is spastic
EMG study | 6th weeks
  Fwave , H reflexElectrophysiological assessment, such as measurement of the reflex activities Spastic muscle: Ankle planter flexor, Knee flexor
Ultrasonography | 6th weeks
  to examine disruptions in the normative architecture of spastic muscles. Muscle length (MFL),Muscle thickness (MT) Muscle pennation angle
Time up and Go | 6th weeks
  To determine fall risk and measure the progress of balance, sit to stand and walking. ≤ 10 seconds = normal. ≤ 20 seconds = good mobility, can go out alone, mobile without gait aid. ≤ 30 seconds = problems, cannot go outside alone, requires gait aid. * A score of ≥ 14 seconds has been shown to indicate high risk of falls.
Burg Balance scale | 6th weeks
  It is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks A score of 56 indicates functional balance. A score of < 45 indicates individuals may be at greater risk of falling.
Functional independence measure | 6th weeks
  The Functional Independence Measure (FIM) is an instrument that was developed as a measure of disability. The FIM's assessment of degree of disability depends on the patient's score in 18 categories, focusing on motor and cognitive function. Each category or item is rated on a 7-point scale (1 = <25% independence; total assistance required, 7 = 100% independence)
Barthal index | 6th weeks
  The Barthel Scale/Index is an ordinal scale used to measure performance in activities of daily living (ADL). It uses ten variables describing ADL and mobility. A higher number is associated with a greater likelihood of being able to live at home with a degree of independence following discharge from hospital. The amount of time and physical assistance required to perform each item are used in determining the assigned value of each item. External factors within the environment affect the score of each item. If adaptations outside the standard home environment are met during assessment, the participant's score will be lower if these conditions are not available.
Rivermead Mobility Index | 6 week
  The Rivermead Mobility Index assesses functional mobility in gait, balance and transfers after stroke. Items receive a score of 0 for a "No" response and 1 for a "Yes" response. Total scores are determined by summing the points for all items. A maximum of 15 points is possible; higher scores indicate better mobility performance. A score of "0" indicates an inability to perform any of the activities on the measure.

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PHD, Principal Investigator — Riphah international university lahore campus
Locations (1):
- Riphah international university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leng Y, Lo WLA, Hu C, Bian R, Xu Z, Shan X, Huang D, Li L. The Effects of Extracorporeal Shock Wave Therapy on Spastic Muscle of the Wrist Joint in Stroke Survivors: Evidence From Neuromechanical Analysis. Front Neurosci. 2021 Jan 21;14:580762. doi: 10.3389/fnins.2020.580762. eCollection 2020. PMID 33551718
- [Background] Carey L, Walsh A, Adikari A, Goodin P, Alahakoon D, De Silva D, Ong KL, Nilsson M, Boyd L. Finding the Intersection of Neuroplasticity, Stroke Recovery, and Learning: Scope and Contributions to Stroke Rehabilitation. Neural Plast. 2019 May 2;2019:5232374. doi: 10.1155/2019/5232374. eCollection 2019. PMID 31191637
- [Background] Arya KN, Verma R, Garg RK, Sharma VP, Agarwal M, Aggarwal GG. Meaningful task-specific training (MTST) for stroke rehabilitation: a randomized controlled trial. Top Stroke Rehabil. 2012 May-Jun;19(3):193-211. doi: 10.1310/tsr1903-193. PMID 22668675
- [Background] Hsu PC, Chang KV, Chiu YH, Wu WT, Ozcakar L. Comparative Effectiveness of Botulinum Toxin Injections and Extracorporeal Shockwave Therapy for Post-Stroke Spasticity: A Systematic Review and Network Meta-Analysis. EClinicalMedicine. 2021 Dec 4;43:101222. doi: 10.1016/j.eclinm.2021.101222. eCollection 2022 Jan. PMID 34927035
- [Background] Mihai EE, Dumitru L, Mihai IV, Berteanu M. Long-Term Efficacy of Extracorporeal Shock Wave Therapy on Lower Limb Post-Stroke Spasticity: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Clin Med. 2020 Dec 29;10(1):86. doi: 10.3390/jcm10010086. PMID 33383655
- [Background] Cabanas-Valdes R, Calvo-Sanz J, Urrutia G, Serra-Llobet P, Perez-Bellmunt A, German-Romero A. The effectiveness of extracorporeal shock wave therapy to reduce lower limb spasticity in stroke patients: a systematic review and meta-analysis. Top Stroke Rehabil. 2020 Mar;27(2):137-157. doi: 10.1080/10749357.2019.1654242. Epub 2019 Nov 11. PMID 31710277
- [Background] Xing Y, Bai Y. A Review of Exercise-Induced Neuroplasticity in Ischemic Stroke: Pathology and Mechanisms. Mol Neurobiol. 2020 Oct;57(10):4218-4231. doi: 10.1007/s12035-020-02021-1. Epub 2020 Jul 20. PMID 32691303
- [Background] Penna LG, Pinheiro JP, Ramalho SHR, Ribeiro CF. Effects of aerobic physical exercise on neuroplasticity after stroke: systematic review. Arq Neuropsiquiatr. 2021 Sep;79(9):832-843. doi: 10.1590/0004-282X-ANP-2020-0551. PMID 34669820
- [Background] Dejong G, Horn SD, Gassaway JA, Slavin MD, Dijkers MP. Toward a taxonomy of rehabilitation interventions: Using an inductive approach to examine the "black box" of rehabilitation. Arch Phys Med Rehabil. 2004 Apr;85(4):678-86. doi: 10.1016/j.apmr.2003.06.033. PMID 15083447
- [Background] Bell ML, Whitehead AL, Julious SA. Guidance for using pilot studies to inform the design of intervention trials with continuous outcomes. Clin Epidemiol. 2018 Jan 18;10:153-157. doi: 10.2147/CLEP.S146397. eCollection 2018. PMID 29403314
- [Background] Yelnik AP, Simon O, Parratte B, Gracies JM. How to clinically assess and treat muscle overactivity in spastic paresis. J Rehabil Med. 2010 Oct;42(9):801-7. doi: 10.2340/16501977-0613. PMID 20878038
- [Background] Rahayu UB, Wibowo S, Setyopranoto I, Hibatullah Romli M. Effectiveness of physiotherapy interventions in brain plasticity, balance and functional ability in stroke survivors: A randomized controlled trial. NeuroRehabilitation. 2020;47(4):463-470. doi: 10.3233/NRE-203210. PMID 33164953
- [Background] Dromerick AW, Geed S, Barth J, Brady K, Giannetti ML, Mitchell A, Edwardson MA, Tan MT, Zhou Y, Newport EL, Edwards DF. Critical Period After Stroke Study (CPASS): A phase II clinical trial testing an optimal time for motor recovery after stroke in humans. Proc Natl Acad Sci U S A. 2021 Sep 28;118(39):e2026676118. doi: 10.1073/pnas.2026676118. PMID 34544853
- [Background] Linder SM, Rosenfeldt AB, Davidson S, Zimmerman N, Penko A, Lee J, Clark C, Alberts JL. Forced, Not Voluntary, Aerobic Exercise Enhances Motor Recovery in Persons With Chronic Stroke. Neurorehabil Neural Repair. 2019 Aug;33(8):681-690. doi: 10.1177/1545968319862557. Epub 2019 Jul 17. PMID 31313626
- [Derived] Afzal B, Noor R, Alghwiri AA, Umar A. Effects of Extracorporeal Shockwave Therapy Combined with Neuroplasticity-Based Training Protocol on Lower Limb Spasticity in Stroke Patients: A Randomized Controlled Trial with Ultrasonography Evaluation. NeuroRehabilitation. 2026 Jan 7:10538135251403026. doi: 10.1177/10538135251403026. Online ahead of print. PMID 41499331